CLINICAL TRIAL: NCT03759301
Title: Efficacy of Growth Hormone Supplementation With Gonadotrophins in IVF/ICSI for Poor Responders; a Randomized Controlled Trial
Brief Title: Efficacy of Growth Hormone Supplementation With Gonadotrophins in IVF/ICSI for Poor Responders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ClinAmygate (Other)
Collaborators: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Emad Roushdy, Director, ClinAmygate
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NRC 0214
Record Dates: First submitted 2018-11-22; First posted 2018-11-29 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Infertility, Female
Keywords: Growth Hormone; IVF/ICSI; Poor Responders
MeSH Terms: conditions — Infertility, Female | interventions — Growth Hormone; cetrorelix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Growth Hormones Somatropin Recombinant (Active Comparator): Growth hormone (Somatropin) 4 IU/day subcutaneous from the 2nd day of the cycle and stopped 1 day before ovum pickup for the treatment group which consists of 70 women.
  Interventions: Drug: Growth Hormones Somatropin Recombinant
- Placebo saline solution (Placebo Comparator): Control group consisting of 70 women who will receive subcutaneous placebo injection in the same dosing as the treatment group
  Interventions: Drug: Placebo saline solution

INTERVENTIONS:
Drug: Growth Hormones Somatropin Recombinant — Growth Hormones Somatropin Recombinant 4 IU/day subcutaneous from the 2nd day of the cycle and stopped 1 day before ovum pickup
  Other Names: Cetrorelix
  Arms: Growth Hormones Somatropin Recombinant
Drug: Placebo saline solution — same volume as growth hormone ampule used
  Other Names: Cetrorelix
  Arms: Placebo saline solution

SUMMARY:
The objective of this study is to assess the effectiveness of adjuvant growth hormone injection during controlled ovarian stimulation, in poor responder women undergoing intracytoplasmic sperm injection (ICSI) procedures.

DETAILED DESCRIPTION:
Infertility is defined as the failure to achieve a clinical pregnancy after 12 months or more of regular unprotected sexual intercourse (and there is no other reason, such as breastfeeding or postpartum amenorrhoea). Primary infertility is infertility in a couple who have never had a child. Secondary infertility is a failure to conceive following a previous pregnancy.

Subfertility, usually defined as the absence of conception after one year of regular intercourse, subfertility is a common problem affecting as many as one in six couples.

According to the European Society of Human Reproduction and Embryology (ESHRE) recommendations, couples with an estimated live birth rate of 40% or higher per year are encouraged to continue aiming for a spontaneous pregnancy .

Treatment methods for infertility may be grouped as medical, complementary and alternative treatments. Some methods may be used in concert with other methods. Drugs may be used for both women and men.

If conservative medical treatments fail to achieve a full term pregnancy, the physician may suggest the patient undergo assisted reproductive fertilization (ART). Methods for ART include artificial insemination (IUI), gamete intrafallopian transfer (GIFT), zygot intrafallopian transfer (ZIFT) or ICSI.

Intracytoplasmic sperm injection (ICSI) is an in vitro fertilization procedure in which a single sperm is injected directly into an oocyte. During the past decade, ICSI has been applied increasingly around the world to alleviate problems of severe male infertility because too few motile and morphologically normal sperm were present in the ejaculate of the male partner.

Although there have been several improvements in techniques of ART during the last three decades clinical pregnancy and live-birth rates remain at approximately 30-40%.

Increasing these rates is desirable for couples undergoing ART, as treatment failure is a source of psychological distress, and the most common cause of drop-out before achieving pregnancy.The most common interventions to improve ART outcome are the use of maximized controlled ovarian stimulation (COS), transference of multiple embryos into the uterus and cryopreservation of surplus oocytes/embryos. However, the first two of these interventions might increase the risk of ovarian hyperstimulation syndrome and multiple pregnancy.

In-vitro fertilization (IVF) protocols are constantly under review in an attempt to decrease hormone (gonadotrophin) requirement, improve follicular recruitment, whilst primarily to increase live birth rates.

Implantation failure is thought to result from impairment of embryo development and/or from abnormal uterine receptivity.

Some protocols have considered the role of growth hormone in IVF. Growth hormone is a biological peptide hormone, synthesized, stored and secreted by somatotroph cells located in the anterior pituitary gland. Growth hormone can be synthetically produced using recombinant DNA technology and is licensed to be used in the human population. There is currently no consensus as to the route, dose or timing of growth hormone administration in IVF protocols.

Poor Ovarian Response (POR) is defined by the Bologna criteria, with an incidence between 9 and 24% of all cycles of IVF, usually it indicates a reduction in follicular response, resulting in a reduced number of retrieved oocytes. It has been recognized that, in order to define the poor response in IVF, at least two of the following three features must be present: (i) advanced maternal age or any other risk factor for POR; (ii) a previous POR; and (iii) an abnormal ovarian reserve test (ORT). Two episodes of POR after maximal stimulation are sufficient to define a patient as poor responder in the absence of advanced maternal age or abnormal ORT. By definition, the term POR refers to the ovarian response, and therefore, one stimulated cycle is considered essential for the diagnosis of POR. However, patients of advanced age with an abnormal ORT may be classified as poor responders since both advanced age and an abnormal ORT may indicate reduced ovarian reserve and act as a surrogate of ovarian stimulation cycle outcome. In this case, the patients should be more properly defined as 'expected poor responder'. If this definition of POR is uniformly adapted as the 'minimal' criteria needed to select patients for future clinical trials, more homogeneous populations will be tested for any new protocols. Finally, by reducing bias caused by spurious POR definitions, it will be possible to compare results and to draw reliable conclusions.

How the intervention might work? The administration of growth hormone may potentiate the effect of exogenous gonadotrophins. Growth hormone is reported to modulate the action of follicular stimulating hormone on granulosa cells by up-regulating the local synthesis of insulin-like growth factor-I (IGF-1). This interest has been stimulated by animal studies which suggest that growth hormone may increase the intra-ovarian production of the IGF-1. IGF-1 displays growth hormone dependence both in-vivo and in-vitro The interaction between growth hormone and IGF-1 is of significance since IGF-1 has been shown to play an important part in ovarian function in both animal and human models. The addition of IGF-1 to gonadotrophins in granulosa cell cultures increased gonadotrophin action on the ovary by several mechanisms including augmentation of aromatase activity, 17 beta-oestradiol and progesterone production and luteinising hormone receptor formation. IGF-1 has also been found to stimulate follicular development, oestrogen production and oocyte maturation.

Improving the outcomes of ICSI by the use of growth hormone adjuvant therapy is important particularly in those women who are considered poor responders. The aim of this study is to establish the role of growth hormone in ICSI.

ELIGIBILITY:
Inclusion Criteria:

* Age: 25 to 38 years old.
* IVF previous poor responders: at least two failed cycles with < five oocytes or abnormal ORT e.g. antimullerian hormone < 1
* Patients with unexplained infertility.
* Normal follicle stimulating hormone (FSH), luteinizing hormone (LH), prolactin and ovarian ultrasound.
* Normal pelvic ultrasound including 3D ultrasound of the uterus with no detected hydrosalpinx.

Exclusion Criteria:

* Refusal to participate in the study
* Patients with known medical disease (e.g. severe hypertension or hepatic disease).
* Altered karyotype in one or both partners.
* History of chronic, autoimmune or metabolic diseases
* Presence of endocrinopathies.

Ages: 25 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 156 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | 3 weeks
  The main outcome is clinical pregnancy per allocated woman, defined as the presence of at least one fetus with heart beat.

SECONDARY OUTCOMES:
E2 levels | Day 1 of COS, the same day of Human Chorionic Gonadotropin (HCG) injection
  Human Chorionic Gonadotropin (HCG) is given to induce triggering of ovulation then ovum pick up is scheduled 36 hour after the injection.
Number of oocytes collected | Day 6 of COS
  Transvaginal ultrasound will be done starting from day 6 of COS for assessment of follicular development and assessment of endometrial thickness, serial E2 measurement will be scheduled to start on day 6 of COS repeating every other day
Metaphase I (MI) and Metaphase II (MII) oocyte number | Day 6 of COS
  Transvaginal ultrasound will be done starting from day 6 of COS for assessment of follicular development and assessment of endometrial thickness, serial E2 measurement will be scheduled to start on day 6 of COS repeating every other day
Number of Pronucleus | Day 6 of COS
  Transvaginal ultrasound will be done starting from day 6 of COS for assessment of follicular development and assessment of endometrial thickness, serial E2 measurement will be scheduled to start on day 6 of COS repeating every other day
Multiple pregnancy | 6 weeks from last period
  Multiple pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Shafeek, MSc, Principal Investigator — Al-Azhar University
Locations (1):
- Al Azhar University Hospitals (Kasr Al-Aini), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sood A, Mohiyiddeen G, Ahmad G, Fitzgerald C, Watson A, Mohiyiddeen L. Growth hormone for in vitro fertilisation (IVF). Cochrane Database Syst Rev. 2021 Nov 22;11(11):CD000099. doi: 10.1002/14651858.CD000099.pub4. PMID 34808697
- [Derived] Mohammad EH, Abou El Serour AG, Mohamed EAH, Abbasy AH, Zaatar M, Rageh KA, Shafeek MM, Issak ER. Efficacy of growth hormone supplementation with ultrashort GnRH antagonist in IVF/ICSI for poor responders; randomized controlled trial. Taiwan J Obstet Gynecol. 2021 Jan;60(1):51-55. doi: 10.1016/j.tjog.2020.10.003. PMID 33495008